CLINICAL TRIAL: NCT03538795
Title: Priming the Brain for Rehabilitation: Brain Stimulation Followed by Constraint-Induced Movement Therapy in Adults With Severe Arm Paresis After Stroke
Brief Title: Brain Stimulation and Rehabilitation for Adults With Chronic, Severe Arm Motor Impairment After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Ran out of funds
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: NIH National Rehabilitation Research Resource to Enhance Clinical Trials (Unknown)
Responsible Party: Principal Investigator, Gitendra Uswatte, Professor of Psychology and Physical Therapy, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-170530008
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Hemiplegia; Hemiparesis
Keywords: stroke; hemiplegia; hemiparesis; arm; upper-extremity; motor impairment; transcranial magnetic stimulation (TMS); brain stimulation; neuroplasticity
MeSH Terms: conditions — Stroke; Hemiplegia; Paresis | interventions — Transcranial Magnetic Stimulation; Constraint Induced Movement Therapy

STUDY DESIGN:
Intervention Model Description: Case series, with a no-treatment control period before the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- iTBS&eCIMT (Experimental): Participants will first receive baseline testing followed by a no-treatment control period. Participants will then be tested again, receive the combination therapy, i.e., iTBS&eCIMT, and then receive post-treatment testing.
  Interventions: Combination Product: iTBS&eCIMT

INTERVENTIONS:
Combination Product: iTBS&eCIMT — All will receive eCIMT+iTBS on an outpatient basis for 4 hours/day for 15 consecutive weekdays. eCIMT will include training of the more-affected arm following shaping principles, restraint of the less-affected arm, and the Transfer Package in combination with NDT techniques to reduce tone so that shaping of movement can be carried out. The Transfer Package is a set of behavioral techniques designed to transfer therapeutic gains from the treatment setting to everyday life. iTBS will be added to prime the areas of the brain that control movement of the more-affected arm so that the responsiveness of that tissue to motor training is enhanced. Treatment sessions will alternate between 10 minute periods of iTBS (which include time for set-up and transition) and 1-hour periods of eCIMT.
  Other Names: CI therapy; TMS; repetitive transcranial magnetic stimulation (rTMS); Constraint-Induced Movement therapy; Transcranial Magnetic Stimulation

SUMMARY:
This pilot study will examine a combination therapy for adults with chronic, severe motor impairment of an arm after stroke. The intervention will combine brain stimulation with physical rehabilitation of the arm on the side of the body more-affected by stroke.

DETAILED DESCRIPTION:
The overarching goal of this program of research is to develop a therapy that produces meaningful and persistent improvements in function of the more-affected arm in stroke survivors with severe, chronic hemiparesis. No treatment with an established evidence base is available now for this large group, who have barely perceptible voluntary movement of the more-affected fingers and wrist. The lab of E. Taub and G. Uswatte has developed an expanded version of Constraint-Induced Movement therapy (CIMT) for this population that has evidence of efficacy for improving use in daily life of the more-affected arm from a case series and small randomized controlled trial (RCT). The original version of CIMT is a form of physical rehabilitation that has evidence of efficacy from multiple RCTs for improving use in daily life of the more-affected arm in adults with mild to moderate hemiparesis after stroke. CIMT has also been shown to produce neuroplastic changes in both grey and white matter structures. Expanded CIMT (eCIMT) combines CIMT with neurodevelopmental techniques (NDT) for managing tone. Studies from by J. Szaflarski and by others suggest that priming CNS tissue for training by electrically stimulating the brain regions that control the target function with excitatory intermittent theta burst stimulation (iTBS) augments the benefits of neurorehabilitation. This pilot study will evaluate the feasibility of combining eCIMT with brain stimulation by iTBS and, on a preliminary basis, will evaluate whether this combination therapy boosts treatment outcomes relative to eCIMT alone.

ELIGIBILITY:
Inclusion Criteria:

* stroke
* > 12 months after stroke onset
* severe hemiparesis of more-affected arm

Exclusion Criteria:

* substantial use of the more-affected arm in daily life
* frailty or insufficient stamina to carry out the requirements of the therapy
* other neurological or musculoskeletal problems, including pain, affecting the more-affected arm
* severe cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gitendra Uswatte, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited from a list of stroke survivors who have contacted our lab but have been excluded from past studies because their motor impairment was too severe. The recruitment period was June 11, 2018 to February 14, 2019.
Groups:
- iTBS&eCIMT: Participants will first receive baseline testing followed by a no-treatment control period. Will then be tested again, receive the combination therapy, i.e., iTBS&eCIMT, and then receive post-treatment testing. Intermittent Theta Burst Stimulation (iTBS) & Expanded Constraint-Induced Movement Therapy (eCIMT): All will receive eCIMT+iTBS on an outpatient basis for 4 hours/day for 15 consecutive weekdays. eCIMT will include training of the more-affected arm following shaping principles, restraint of the less-affected arm, and the Transfer Package in combination with neurodevelopmental techniques (NDT) techniques to reduce tone so that shaping of movement can be carried out. The Transfer Package is a set of behavioral techniques designed to transfer therapeutic gains from the treatment setting to everyday life. iTBS will be added to prime the areas of the brain that control movement of the more-affected arm so that the responsiveness of that tissue to motor training is enhanced.
Period: Overall Study
Arm/Group | iTBS&eCIMT
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- iTBS&eCIMT: Participants will first receive baseline testing followed by a no-treatment control period. Participants will then be tested again, receive the combination therapy, i.e., iTBS&eCIMT, and then receive post-treatment testing. iTBS&eCIMT: All will receive eCIMT+iTBS on an outpatient basis for 4 hours/day for 15 consecutive weekdays. eCIMT will include training of the more-affected arm following shaping principles, restraint of the less-affected arm, and the Transfer Package in combination with NDT techniques to reduce tone so that shaping of movement can be carried out. The Transfer Package is a set of behavioral techniques designed to transfer therapeutic gains from the treatment setting to everyday life. iTBS will be added to prime the areas of the brain that control movement of the more-affected arm so that the responsiveness of that tissue to motor training is enhanced. Treatment sessions will alternate between 10 minute periods of iTBS (which include time for set-up and transition)
Arm/Group | iTBS&eCIMT
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Motor Activity Log (MAL)
Description: Structured interview that assesses use of the more-affected arm in daily life. Scale range is 0 (no use of the more-affected arm) to 5 (use that is as good before stroke). Higher scores are better. Score reported is change from Day 0 to Day 42.
Time Frame: Change from Day 0 to Day 42
Measure: Mean (Standard Deviation); unit: units on a scale, range = 0-5
Groups:
- iTBS&eCIMT: Participants will first receive baseline testing followed by a no-treatment control period. Participants will then be tested again, receive the combination therapy, i.e., iTBS&eCIMT, and then receive post-treatment testing. iTBS&eCIMT: All will receive eCIMT+iTBS on an outpatient basis for 4 hours/day for 15 consecutive weekdays. eCIMT will include training of the more-affected arm following shaping principles, restraint of the less-affected arm, and the Transfer Package in combination with NDT techniques to reduce tone so that shaping of movement can be carried out. The Transfer Package is a set of behavioral techniques designed to transfer therapeutic gains from the treatment setting to everyday life. iTBS will be added to prime the areas of the brain that control movement of the more-affected arm so that the responsiveness of that tissue to motor training is enhanced. Treatment sessions will alternate between 10 minute periods of iTBS and 1-hour periods of eCIMT.
Arm/Group | iTBS&eCIMT
Number analyzed (Participants) | 3
units on a scale, range = 0-5 | 1.8 (0.6)

2. Secondary Outcome: Wolf Motor Function Test (WMFT)
Description: Laboratory motor performance test that assesses motor capacity of the more-affected arm. Scale range is 0 to infinite. Higher scores are better.
Time Frame: Change from Day 0 to Day 42
Population: Study terminated early due to lack of funds. No funds available to score this test for the 3 participants who completed the study. Unable to analyze due to smaller than projected sample size.
Arm/Group | iTBS&eCIMT
Number analyzed (Participants) | 0

3. Secondary Outcome: Canadian Occupational Performance Measure (COPM)
Description: Structured interview that assesses use of the arms in daily life
Time Frame: Change from Day 0 to Day 42
Population: Study terminated early due to lack of funds. No funds available to score this test for the 3 participants who completed study. Unable to analyze outcome due to smaller than projected sample size.
Arm/Group | iTBS&eCIMT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 42 days
Description: Selected, anticipated medical problems in the target population, i.e, stroke, were assessed either as part of the outcome testing or trainers and testers regularly asked about the presence of symptoms of interest.
Arm/Group | iTBS&eCIMT
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTBS&eCIMT (N=3)
Elevated blood pressure (Vascular disorders) | 1 (1) — Not related to participation.
Pain (Nervous system disorders) | 1 (3) — Related to study but anticipated. Problems with pain are a feature of stroke.
Depressive symptoms (Psychiatric disorders) | 1 (1) — Not related to study. Depressive symptoms are a feature of stroke. Did not meet criteria for major depressive disorder. Denied suicidal ideation.
Lethargy (Metabolism and nutrition disorders) | 1 (1) — Not related to study. Side effect of medication prescribed by participant's personal physician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT03538795/Prot_SAP_000.pdf